CLINICAL TRIAL: NCT03638960
Title: Interscalene Single Shot With Plain Bupivacaine Versus Liposomal Bupivacaine for Arthroscopic Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Gligor Gucev, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APP-18-01917
Record Dates: First submitted 2018-08-08; First posted 2018-08-20 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2021-09

CONDITIONS: Shoulder Pain; Postoperative Pain
Keywords: peripheral nerve block; interscalene; arthroscopic shoulder surgery; liposomal bupivacaine
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: The investigators plan to perform a double blinded randomized control study. Patients will be randomly assigned to either group A or group B. Patients in group A will receive a bolus injection with 20 mL of 0.5% bupivacaine. Group B will receive 10 mL of 133 mg of liposomal bupivacaine mixed with 10 mL 0.5% bupivacaine.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and data collectors are unaware of which group the patient belongs to. The anesthesiologist performing the nerve block will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Active Comparator): Patients in group A will receive a bolus injection with 20 mL of 0.5% bupivacaine.
  Interventions: Drug: Bupivacaine Hydrochloride
- Liposomal bupivacaine (Experimental): Group B will receive 10 mL of 133 mg of liposomal bupivacaine mixed with 10 mL 0.5% bupivacaine.
  Interventions: Drug: Bupivacaine liposome

INTERVENTIONS:
Drug: Bupivacaine liposome — The investigators will perform an ultrasound-guided interscalene peripheral nerve block with either liposomal bupivacaine prior to the patient receiving surgery.
  Other Names: peripheral nerve block
  Arms: Liposomal bupivacaine
Drug: Bupivacaine Hydrochloride — The investigators will perform an ultrasound-guided interscalene peripheral nerve block with either plain bupivacaine prior to the patient receiving surgery.
  Other Names: peripheral nerve block
  Arms: Bupivacaine

SUMMARY:
The investigators will be comparing pain scores and opioid use in patients receiving interscalene peripheral blocks with plain bupivacaine versus those receiving liposomal bupivacaine. Liposomal bupivacaine is described as releasing local anesthetic up to 72 hours after its injection; therefore if liposomal bupivacaine can provide extended pain relief compared to plain bupivacaine, the investigators can consider using it as our primary local anesthetic. As secondary outcomes, the investigators will also be looking at difference in functional status and long-term differences between the two local anesthetics.

DETAILED DESCRIPTION:
Background:

The current standard of care for patients at the investigators' institution is to perform an interscalene peripheral nerve block for patients receiving arthroscopic shoulder surgery surgery as it is an effective opioid-free alternative for post-operative pain control. The investigators in the past perform both single shot injections and place catheter based on patient and surgical preferences. Catheters have shown to have extended benefit throughout the perioperative period, including lower pain scores, reduced analgesics and improved sleep. However, the negatives of catheters include the placement of a foreign body, increased time to perform the procedure, interference in surgical field and increased cost of catheter equipment and local anesthetic pump and premature catheter dislodgement. Therefore, pros and cons of deciding between placing a single shot injecting versus catheter has to be considered individually for each case.

Liposomal bupivacaine due to its liposomal outer layers, releases bupivacaine over a longer period of time than plain bupivacaine. A pharmacokinetic study showed the terminal half-life of bupivacaine to be 131 ± 58 minutes versus 1294 ± 860 minutes for liposomal bupivacaine.

In a recent study comparing liposomal bupivacaine to placebo for interscalene peripheral nerve blocks, patients receiving liposomal bupivacaine had significantly lower pain scores over 48 hours and received less opioid over 72 hours[6]. Therefore, if a single shot injection with liposomal bupivacaine can provide longer pain relief than plain bupivacaine, it makes the decision to perform single shot interscalene peripheral nerve blocks easier.

Study Objectives The investigators would like to study whether an interscalene peripheral block injection with liposomal bupivacaine provides superior pain control compared to an interscalene single shot with plain bupivacaine. The investigators will be looking at average daily pain scores, highest daily visual analog scale (VAS) pain scores at rest and with movement, total daily opioid consumption from immediately post-operative to 7 days post-operative, and functionality with physical therapy. The investigators will also plan to follow these patients 6 month and 12 months post-operative to determine whether there is any difference in incidence of persistent post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* medically optimized patients that will undergo an elective surgery for arthroscopic shoulder surgery

Exclusion Criteria:

* under 18 years pregnant or breast-feeding, non-English speaking, have renal or hepatic dysfunction, history of chronic opioid use, receiving worker's compensation, smoker, receiving capsular release, respiratory compromise or BMI < 18 or > 35 or allergy to local anesthetics or opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Average worst pain score with movement over 3 days | 3 days post-operative
  The investigators will assess the patients worst pain score each day with movement up to 3 days post-operative. Pain will be assessed using the visual analog scale (VAS) with 0 indicating no pain and 10 indicating worst pain.

SECONDARY OUTCOMES:
Average worst pain score with movement over 7 days | 7 days post-operative
  The investigators will assess the patients worst pain score each day with movement up to 7 days post-operative. Pain will be assessed using the visual analog scale (VAS) with 0 indicating no pain and 10 indicating worst pain.
Total opioid use over 3 days | 3 days post-operative
  The investigators will calculate opioid use by recording opioid consumption from patient responses. The total consumption will be converted to morphine equivalents.
Total opioid use over 7 days | 7 days post-operative
  The investigators will calculate opioid use by recording opioid consumption from patient responses. The total consumption will be converted to morphine equivalents.
Functional Assessment with Physical Therapy | Up to 1 month post-operative
  Physical therapy function will be assessed using the Shoulder Function Classification System (SFCS). Patients will receive a score between 0 (poor functional status) - 100 (full function).
Risk of persistent post-operative pain at 6 months & 12 months | 6 months, 12 months
  Patients will be interviewed with the Brief Pain Inventory (BPI) at 6 and 12 months post-operative to assess persistent pain.
Adverse events | 7 days
  This includes nausea/vomiting, nerve injury, local anesthetic toxicity, unexpected readmission or emergency room visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho CH, Song KS, Min BW, Jung GH, Lee YK, Shin HK. Efficacy of interscalene block combined with multimodal pain control for postoperative analgesia after rotator cuff repair. Knee Surg Sports Traumatol Arthrosc. 2015 Feb;23(2):542-7. doi: 10.1007/s00167-012-2272-3. Epub 2012 Oct 30. PMID 23108685
- [Background] Liu XN, Noh YM, Yang CJ, Kim JU, Chung MH, Noh KC. Effects of a Single-Dose Interscalene Block on Pain and Stress Biomarkers in Patients Undergoing Arthroscopic Rotator Cuff Repair: A Randomized Controlled Trial. Arthroscopy. 2017 May;33(5):918-926. doi: 10.1016/j.arthro.2016.09.018. Epub 2016 Dec 14. PMID 27988164
- [Background] Salviz EA, Xu D, Frulla A, Kwofie K, Shastri U, Chen J, Shariat AN, Littwin S, Lin E, Choi J, Hobeika P, Hadzic A. Continuous interscalene block in patients having outpatient rotator cuff repair surgery: a prospective randomized trial. Anesth Analg. 2013 Dec;117(6):1485-92. doi: 10.1213/01.ane.0000436607.40643.0a. PMID 24257398
- [Background] Malik T, Mass D, Cohn S. Postoperative Analgesia in a Prolonged Continuous Interscalene Block Versus Single-Shot Block in Outpatient Arthroscopic Rotator Cuff Repair: A Prospective Randomized Study. Arthroscopy. 2016 Aug;32(8):1544-1550.e1. doi: 10.1016/j.arthro.2016.01.044. Epub 2016 Apr 20. PMID 27107906
- [Background] Davidson EM, Barenholz Y, Cohen R, Haroutiunian S, Kagan L, Ginosar Y. High-dose bupivacaine remotely loaded into multivesicular liposomes demonstrates slow drug release without systemic toxic plasma concentrations after subcutaneous administration in humans. Anesth Analg. 2010 Apr 1;110(4):1018-23. doi: 10.1213/ANE.0b013e3181d26d2a. PMID 20357145
- [Background] Keller S, Bann CM, Dodd SL, Schein J, Mendoza TR, Cleeland CS. Validity of the brief pain inventory for use in documenting the outcomes of patients with noncancer pain. Clin J Pain. 2004 Sep-Oct;20(5):309-18. doi: 10.1097/00002508-200409000-00005. PMID 15322437
- [Background] Pacira Pharmaceuticals, I., Efficacy, Safety, and Pharmacokinetics of Brachial Plexus Block With EXPAREL in Shoulder Surgery. 2016.